CLINICAL TRIAL: NCT01957761
Title: Molecular Epidemiologic Survey and Risk Factor Assessment of Clostridium Difficile Infections in Children: A Focus on Recurrent and Community-associated Infections
Brief Title: Molecular Epidemiology of Clostridium Difficile Infections in Children
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: Merck MISP 50366
Record Dates: First submitted 2012-11-19; First posted 2013-10-08 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2013-10

CONDITIONS: Clostridium Difficile Infections
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clostridium difficile infection

SUMMARY:
Objectives:

1. Describe the molecular epidemiology of Clostridium Difficile infection in children in the Chicago area.
2. Determine the clinical spectrum and risk factors for Clostridium Difficile infection secondary to particular endemic strains in children.
3. Define the risk factors for recurrent and community-associated Clostridium Difficile infection in children.

ELIGIBILITY:
Inclusion Criteria:

* Clostridium Difficile infection

Exclusion Criteria:

* Age < 1 year
* Age > 18 years

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Clostridium Difficile infection
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clostridium Difficile Infection: All patients with CDI between 12/2012 and 12/2013 were retrospectively reviewed.
Period: Overall Study
Arm/Group | Clostridium Difficile Infection
Started | 189
Completed | 189
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clostridium Difficile Infection
Number analyzed (Participants) | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 176
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 9 [1 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 111
Region of Enrollment [Number; unit: participants]
  United States | 189
Number of cases of BI/NAP1/027 [Number; unit: cases] | 3

OUTCOME MEASURES:

1. Primary Outcome: Clostridium Difficile Infections Strain Type Based on Restriction Endonuclease Analysis
Description: Stool samples taken from patients with Clostridium Difficile Infections infection at the time of diagnosis will be assessed by restriction endonuclease analysis to determine strain type. In order to study the relationship between strain type and outcome of their infection (e.g, treatment failure, recurrence, complication of illness), patients will be followed throughout their illness and for 8 weeks after developing their infection.
Time Frame: On day 1 of diagnosis of Clostridium difficile infection
Measure: Number; unit: cases of BI/NAP1/027
Arm/Group | Clostridium Difficile Infection
Number analyzed (Participants) | 189
cases of BI/NAP1/027 | 3

ADVERSE EVENTS:
Arm/Group | Clostridium Difficile Infection
Serious Adverse Events (participants affected / at risk) | 0/189
Other Adverse Events (participants affected / at risk) | 0/189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No